CLINICAL TRIAL: NCT00335283
Title: Randomized Placebo-Controlled Trial of BID Lansoprazole in Isolated Chronic Post Nasal Drip
Brief Title: Efficacy of Lansoprazole in Chronic Post Nasal Drip
Acronym: PND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: TAP Pharmaceutical Products Inc. (Industry)
Responsible Party: Principal Investigator, Michael Vaezi, Medical Director, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 051169
Record Dates: First submitted 2006-06-07; First posted 2006-06-09 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-06

CONDITIONS: Larynx Disease
MeSH Terms: conditions — Laryngeal Diseases | interventions — Lansoprazole; Hydrogen-Ion Concentration; Manometry

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lansoprazole (Active Comparator)
  Interventions: Drug: Lansoprazole Tablet; Procedure: PH and impedence testing; Procedure: manometry; Drug: lansoprazole
- Sugar Pill (Placebo Comparator)
  Interventions: Procedure: PH and impedence testing; Procedure: manometry; Drug: placebo

INTERVENTIONS:
Drug: Lansoprazole Tablet — 40 mg bid x 16 weeks
  Other Names: prevacid
  Arms: Lansoprazole
Procedure: PH and impedence testing — 24 hour ph monitoring
Procedure: manometry — done prior to pH probe to measure length of esophagus
Drug: lansoprazole — 40mg bid
  Arms: Lansoprazole
Drug: placebo — one tablet bid
  Arms: Sugar Pill

SUMMARY:
The purpose of this study is to determine whether aggressive acid suppression with Lansoprazole is effective in the treatment of post nasal drip, and also assess the predictors of response based on clinical and physiologic parameters.

DETAILED DESCRIPTION:
Postnasal drip (PND) is a common complaint that brings patients to the attention of their primary care physicians. It is also one of the most common reasons for patients to seek care from otolaryngologists. Traditionally, PND has been considered and treated as a symptom of sinonasal pathology. It has also been shown, along with Gastroesophageal reflux disease (GERD) and asthma, to be a major contributor to the development of chronic cough. PND refractory to treatment aimed at sinonasal disease is sometimes treated with anti-GERD therapy. This treatment modality is based on clinical experience. To date, there are no studies in the literature to support a causal relationship between PND and extraesophageal reflux (EER). In a case control study of patients with and without esophagitis El-Serag et al reported a significant association (odds ratio 1.6, 95%CI 1.4-1.8) between sinusitis and GERD. A later study by Ulualp et al in 11 CT confirmed cases of chronic sinusitis resistant to therapy with conventional sinus therapies they found a significantly higher prevalence of hypopharyngeal acid exposure in the sinusitis group than controls. Recently, in an open label prospective pilot trial, DiBaise et al treated 11 patients with sinusitis and 19 GERD patients with omeprazole 20mg bid for 3-months. 9/11 sinusitis patients were found to have GERD by pH monitoring and there was moderate (25-89%) improvement in the sinus symptoms in the omeprazole treated group. However, there are currently no placebo-controlled trials assessing efficacy of PPI's in patients with PND.

ELIGIBILITY:
Inclusion Criteria:

* Negative RAST inhalant allergy panel OR negative skin testing (Group A)
* Positive RAST or Positive skin testing AND insufficient response to all of the following: (Group B)

  * Allergen avoidance
  * Topical nasal steroids
  * Allergy shots if indicated
  * Antihistamines
  * Negative CT sinuses (coronal)
  * < 4mm of mucosal thickening and < 3 sinus sites
  * Absence of air-fluid levels
  * Negative anterior rhinoscopy
  * Absence of pus, crusts on mucosal surfaces

Exclusion Criteria:

* Age < 18
* Pregnancy, confirmed by urine pregnancy test at day of randomization
* Ciliary dyskinesia
* Immune deficiency
* Cystic fibrosis
* Diagnosis of acute sinusitis or chronic RS (AAO-HNS)
* Active use of topical decongestant
* Use of PPI within the last 30 days
* Previous fundoplication
* Uncontrolled thyroid disease
* Isolated chronic cough without the symptom of post nasal drip

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Vaezi, MD PhD MS, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Vanderbilt Digestive Disease Clinic, TVC, Room 1660, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The PI and/or study coordinator or other GI research nurses will meet with the patients referred by Vanderbilt's Asthma, Sinus and Allergy Program. The patients will be given the consent form to read, the document will be reviewed, and all questions will be answered.
Groups:
- Lansoprazole: 40 mg twice a day
- Placebo (Sugar Pill): one tablet twice a day
Period: Overall Study
Arm/Group | Lansoprazole | Placebo (Sugar Pill)
Started | 36 | 39
Completed | 30 | 34
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lansoprazole | Placebo (Sugar Pill) | Total
Number analyzed (Participants) | 36 | 39 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 36 | 69
  >=65 years | 3 | 3 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 46 (15) | 45 (13) | 45 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 26 | 56
  Male | 6 | 13 | 19
Region of Enrollment [Number; unit: participants]
  United States | 36 | 39 | 75

OUTCOME MEASURES:

1. Primary Outcome: Post Nasal Drainage Symptom Response
Description: The primary outcome measure was postnasal drainage symptom response measured by using a visual analogue scale. At 8 and 16 weeks, a horizontal symptoms scale from 0% (no change) to 100% (symptoms completely resolved) was presented to participants to assess improvement in postnasal drainage symptoms.
Time Frame: 8 and 16 weeks
Population: Analysis was performed per the protocol. At the completion of the study, all data were analyzed by the department of statistics and epidemiologyfor the primary outcome of interest, which was response rate for both lansoprazole and placebo. Univariate and multivariate analyses was performed on the collected data.
Measure: Median (Inter-Quartile Range); unit: Scores on a Scale
Arm/Group | Lansoprazole | Placebo (Sugar Pill)
Number analyzed (Participants) | 30 | 34
Scores on a Scale
  8 week | 55 [12.5 to 80] | 3.5 [0 to 53.8]
  16 week | 50 [10 to 72] | 5 [0 to 40]
Statistical Analysis 1: Comparison: Lansoprazole vs Placebo (Sugar Pill); This applies to the 8 week treatment effect. A sample size of 33 patients in treated arm was considered sufficient to detect a difference of 35% between groups, assuming a lansoprazole treatment response of 70% and a placebo response of 35% with an alpha level of .05 and 90% power. A total of 75 patienst was considered an adequate sample size to allow for a 10% dropout rate; Test type: Superiority or Other; p = .01, Regression, Logistic; Odds Ratio, log = 3.12, 95% CI 2-sided [1.28 to 7.59]
Statistical Analysis 2: Comparison: Lansoprazole vs Placebo (Sugar Pill); This applies to the 16 week treatment affect. A sample size of 33 patients in treated arm was considered sufficient to detect a difference of 35% between groups, assuming a lansoprazole treatment response of 70% and a placebo response of 35% with an alpha level of .05 and 90% power. A total of 75 patienst was considered an adequate sample size to allow for a 10% dropout rate; Test type: Superiority or Other; p = .006, Regression, Logistic; Odds Ratio, log = 3.5, 95% CI 2-sided [1.41 to 8.67]

2. Secondary Outcome: Rhinosinusitis Outcome Measure(RSOM-31)
Description: RSOM-31 includes 31 questions combined into a total score ranging from 0 to 155 with higher scores representing greater disease burden. Values are based on patient report.
Time Frame: Baseline, 8 weeks, and 16 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a Scale
Arm/Group | Lansoprazole | Placebo (Sugar Pill)
Number analyzed (Participants) | 30 | 34
Scores on a Scale
  Baseline | 63 [50 to 93] | 51 [38 to 69]
  8 weeks | 40 [23 to 65] | 36 [20 to 60]
  16 weeks | 35 [21 to 61] | 35 [23 to 55]
Statistical Analysis 1: Comparison: Lansoprazole vs Placebo (Sugar Pill); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .97, Regression, Logistic; Odds Ratio, log = 1.01, 95% CI 2-sided [0.38 to 2.70]
Statistical Analysis 2: Comparison: Lansoprazole vs Placebo (Sugar Pill); This applies to the 16 week treatment effect. A sample size of 33 patients in treated arm was considered sufficient to detect a difference of 35% between groups, assuming a lansoprazole treatment response of 70% and a placebo response of 35% with an alpha level of .05 and 90% power. A total of 75 patienst was considered an adequate sample size to allow for a 10% dropout rate; Test type: Superiority or Other; p = .84, Regression, Logistic; Odds Ratio, log = 1.11, 95% CI 2-sided [0.40 to 3.06]

3. Secondary Outcome: Sino Nasal Outcome Test (SNOT-20)
Description: SNOT-20 includes 20 questions combined into a total score ranging from 0 to 100 with higher numbers representing greater rhinosinusitis health burden and represents patient-reported symptom severity.
Time Frame: Baseline, 8 weeks and 16 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a Scale
Arm/Group | Lansoprazole | Placebo (Sugar Pill)
Number analyzed (Participants) | 30 | 34
Scores on a Scale
  Baseline | 36 [31 to 52] | 35 [31 to 45]
  8 weeks | 25 [17 to 35] | 32 [17 to 39]
  16 weeks | 20 [19 to 40] | 27 [16 to 38]
Statistical Analysis 1: Comparison: Lansoprazole vs Placebo (Sugar Pill); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .06, Regression, Logistic; Odds Ratio, log = 2.44, 95% CI 2-sided [.95 to 6.31]
Statistical Analysis 2: Comparison: Lansoprazole vs Placebo (Sugar Pill); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = .007, Regression, Logistic; Odds Ratio, log = 4.51, 95% CI 2-sided [1.5 to 13.6]

4. Secondary Outcome: Quality of Life Questionnaire (QOLRAD)
Description: The patient-reported QOLRAD consists of 25 questions combined into a total score ranging from 25 to 175 with higher numbers representing better quality of life.
Time Frame: Baseline, 8 weeks and 16 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a Scale
Arm/Group | Lansoprazole | Placebo (Sugar Pill)
Number analyzed (Participants) | 30 | 34
Scores on a Scale
  Baseline | 155 [126 to 169] | 160 [142 to 170]
  8 weeks | 174 [157 to 175] | 155 [148 to 170]
  16 weeks | 173 [158 to 174] | 160 [146 to 172]
Statistical Analysis 1: Comparison: Lansoprazole vs Placebo (Sugar Pill); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .006, Regression, Logistic; Odds Ratio, log = 5.17, 95% CI 2-sided [2.02 to 13.2]
Statistical Analysis 2: Comparison: Lansoprazole vs Placebo (Sugar Pill); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = .001, Regression, Logistic; Odds Ratio, log = 5.31, 95% CI 2-sided [1.97 to 14.3]

ADVERSE EVENTS:
Arm/Group | Lansoprazole | Placebo (Sugar Pill)
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/39
Other Adverse Events (participants affected / at risk) | 0/36 | 0/39

LIMITATIONS AND CAVEATS:
Sample size of 75 participants is small. Lack of an objective measure of postnasal drainage limited the study outcome to be symptom based.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No